CLINICAL TRIAL: NCT00289627
Title: A Multi-Center Single Arm Phase II Study of MDX-010 (BMS-734016) Monotherapy in Patients With Previously Treated Unresectable Stage III or IV Melanoma
Brief Title: A Single Arm Study of Ipilimumab Monotherapy in Patients With Previously Treated Unresectable Stage III or IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Medarex (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-008
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Melanoma
Keywords: Previously treated melanoma; Unresectable Stage III; Stage IV
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

ARMS (1):
- ipilimumab (MDX-010, BMS-734016) (Experimental)
  Interventions: Drug: ipilimumab (MDX-010, BMS-734016)

INTERVENTIONS:
Drug: ipilimumab (MDX-010, BMS-734016) — IV solution, IV, 10 mg/kg, Q 3 wks for 12 wks then Q 12 wks, 48+ weeks depending on response.

SUMMARY:
The purpose of this clinical research study is to evaluate the Best Overall Response Rate (BORR), (as per modified WHO criteria) in patients with previously treated melanoma-Stage III (unresectable) or Stage IV melanoma receiving 10 mg/kg of ipilimumab. The safety of this product will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously treated Stage III (unresectable)or Stage IV melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2006-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Evaluate BORR in patients with previously treated Stage III (unresectable) or Stage IV melanoma receiving ipilimumab.

SECONDARY OUTCOMES:
estimate disease control rate
estimate progression free survival rate at Week 12
estimate PFS
estimate overall survival
estimate survival rate at one year
estimate duration of BOR
evaluate proportion of patients whose duration of response is >=24 weeks
estimate time to BOR
evaluate safety profile of ipilimumab during the induction and maintenance phases
evaluate health-related quality of life
obtain PK sample for population PK analysis

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (53):
- United States (14):
  - Little Rock, Arkansas
  - San Francisco, California
  - Santa Monica, California
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Goshen, Indiana
  - Hazard, Kentucky
  - Albuquerque, New Mexico
  - New York, New York
  - Portland, Oregon
  - Greenville, South Carolina
  - Knoxville, Tennessee
  - Dallas, Texas
  - Charlottesvillle, Virginia
- Austria (3):
  - Local Institution, Salzburg
  - Local Institution, Vienna
  - Local Institution, Wels
- Local Institution, Turku, Finland
- Italy (7):
  - Local Institution, Genova
  - Local Institution, Meldola
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Siena
  - Local Institution, Torino
- Local Institution, Oslo, Norway
- Poland (3):
  - Local Institution, Lodz
  - Local Institution, Poznan
  - Local Institution, Wroclaw
- Russia (9):
  - Local Institution, Barnaul
  - Local Institution, Moscow
  - Local Institution, Murmansk
  - Local Institution, Ryazan
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
  - Local Institution, Stavropol
  - Local Institution, Veliky Novgorod
  - Local Institution, Voronezh
- Spain (5):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Málaga
  - Local Institution, Santa Cruz de Tenerife
  - Local Institution, Valencia
- Sweden (4):
  - Local Institution, Gothenburg
  - Local Institution, Lund
  - Local Institution, Stockholm
  - Local Institution, Uppsala
- Ukraine (6):
  - Local Institution, Cherkassy
  - Local Institution, Dnipropetrovsk
  - Local Institution, Kiev
  - Local Institution, Lviv
  - Local Institution, Sumy
  - Local Institution, Uzhhorod

REFERENCES:
- [Derived] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295
- [Derived] Di Giacomo AM, Danielli R, Guidoboni M, Calabro L, Carlucci D, Miracco C, Volterrani L, Mazzei MA, Biagioli M, Altomonte M, Maio M. Therapeutic efficacy of ipilimumab, an anti-CTLA-4 monoclonal antibody, in patients with metastatic melanoma unresponsive to prior systemic treatments: clinical and immunological evidence from three patient cases. Cancer Immunol Immunother. 2009 Aug;58(8):1297-306. doi: 10.1007/s00262-008-0642-y. Epub 2009 Jan 13. PMID 19139884
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx